CLINICAL TRIAL: NCT07104045
Title: Effect of Reduced Light Color Temperature on Postpartum Mothers' Well-being, Breastfeeding Motivation, and Psychological Well-being After Cesarean Section: A Randomized Placebo-controlled Trial
Brief Title: Effect of Reduced Light Color Temperature on Postpartum Mothers' Well-being, Breastfeeding Motivation, and Psychological Well-being After Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 121212
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Light Color Temperature

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Reduced light color temperature
  Interventions: Other: Reduced light color temperature
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: Reduced light color temperature — reduced light color temperature on postpartum mothers' well-being, breastfeeding motivation, and psychological well-being after a cesarean section
  Arms: Intervention group

SUMMARY:
The aim of this study is to determine the effects of reduced light color temperature on postpartum mothers' well-being, breastfeeding motivation, and psychological well-being after cesarean section. Method: This study is a randomized controlled experimental study conducted with 80 postpartum mothers. Data are collected using a Personal Information Form, the Well-being Scale (HS), the Psychological Well-being Scale (PWB), and the Breastfeeding Motivation Scale (BMS).

ELIGIBILITY:
Inclusion Criteria:

* being in the postpartum process

Exclusion Criteria:

* having communication problems

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 80 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
the Well-being Scale | 12 hours
  Well being
the Peace Scale | 12 hours
  peaces
Breastfeeding Motivation Scale | 12 hours
  Breastfeeding Motivation

IPD SHARING:
Plan to Share IPD: No